CLINICAL TRIAL: NCT03979365
Title: A Prospective, Randomized, Multicenter, Open-Label, Pilot Study to Investigate Medication Adherence & Patient Reported Symptom Occurrence & Interference w/ Daily Life Comparing Envarsus XR® & Immediate Release Tacrolimus in Adult Renal Transplant Recipients (SIMPLE)
Brief Title: Envarsus XR Compared to Immediate Release Tacrolimus
Acronym: SIMPLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Mark Stegall, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-002678
Record Dates: First submitted 2019-05-22; First posted 2019-06-07 (Actual); Results first posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Kidney Transplant Recipients
Keywords: tacrolimus; envarsus xr; renal transplant; kidney transplant
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tacrolimus twice-daily (Active Comparator): Subjects assigned to this arm will take tacrolimus two times daily by mouth, at the clinically prescribed dose.
  Interventions: Drug: Tacrolimus twice daily
- Envarsus XR (Active Comparator): Subjects assigned to this arm will take Envarsus XR one time daily by mouth, at the clinically prescribed dose.
  Interventions: Drug: Envarsus XR

INTERVENTIONS:
Drug: Envarsus XR — Once daily Envarsus XR
  Arms: Envarsus XR
Drug: Tacrolimus twice daily — Twice daily tacrolimus
  Arms: Tacrolimus twice-daily

SUMMARY:
The purpose of this study is to compare once-daily tacrolimus extended-release (Envarsus XR®) to twice-daily immediate release tacrolimus to find out if people taking tacrolimus extended release (Envarsus XR®) report fewer side effects, increased medication compliance and higher scores on quality of life assessments compared to people taking twice daily tacrolimus immediate release.

DETAILED DESCRIPTION:
Despite improvement in short-term graft outcomes in organ transplant, transplant patients still have to take on complex medication regimens to achieve current results. Adherence to these complex medications is an important problem in light of the potential risk of acute and chronic rejection and the associated burden of increased hospitalization, cost, and diminished quality of life that results from missed doses and poor overall drug taking. Part of the diminished quality of life is also tied to the bothersome symptoms patient feel after transplant. Most patients experience symptoms that relate to either the overall transplant immunosuppression or medication specific side effects. In the BENEFIT and BENEFIT-EXT trials, >60% of patients reported tiredness and lack of energy as an issue. Sleep problems, mood swings, restlessness, anxiety, depression, and concentration and memory difficulties appeared in approximately 50-60% of patients. In addition to these symptoms, >38% patients also reported numerous others side effects that have been strongly associated with calcineurin-inhibitors such as tacrolimus that include dizziness, muscle cramps, trembling hands, tingling in hands and feet, and headache.

The investigators hypothesize that the use of once-daily Envarsus XR® could decrease some transplant- and tacrolimus-related adverse symptoms and potentially lead to improvement in quality of life and medication adherence when compared to twice-daily tacrolimus. In order to assess this hypothesis, a prospective, multi-center, randomized, open-label, pilot study to investigate medication adherence and patient reported symptom occurrence and interference with daily life comparing once-daily Envarsus XR® and twice-daily immediate release tacrolimus in adult renal transplant recipients (SIMPLE) is being proposed.

ELIGIBILITY:
Inclusion Criteria:

* Patient is an adult (18 years of age or older).
* Treatment with Envarsus XR® or immediate-release, twice-daily tacrolimus has been indicated by patient's transplant care team.
* Patient is a recipient of a deceased or living donor kidney transplant.
* Patient is able to comply with study procedures for the entire length of the study.
* Patient has been informed about the study survey and has signed an informed consent form.

Exclusion Criteria:

* Patient is unable or unwilling to complete study patient reported outcome questionnaires.
* Patient is currently receiving azathioprine
* Patient is currently receiving an mTOR inhibitor (sirolimus, everolimus)
* Patient is currently receiving an belatacept
* Patient has received investigational immunosuppression 1 month prior to transplant or post-transplant
* Patient is in a setting where a professional care taker is responsible for dispensing subject's medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stegall, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 28 subjects withdrew prior to randomization.
Groups:
- Tacrolimus Twice-daily: Subjects assigned to this arm took tacrolimus two times daily by mouth, at the clinically prescribed dose.
  Tacrolimus twice daily: Twice daily tacrolimus
- Envarsus XR: Subjects assigned to this arm took Envarsus XR one time daily by mouth, at the clinically prescribed dose.
  Envarsus XR: Once daily Envarsus XR
Period: Overall Study
Arm/Group | Tacrolimus Twice-daily | Envarsus XR
Started | 109 | 124
Completed | 108 | 117
Not Completed | 1 | 7
Not completed — Death | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Drug Conversion | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tacrolimus Twice-daily | Envarsus XR | Total
Number analyzed (Participants) | 109 | 124 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.97 (13.38) | 53.91 (14.77) | 54.95 (14.09)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 45 | 46 | 91
  Male | 64 | 77 | 141
  Unknown | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 5
  White | 91 | 86 | 177
  African American or Black | 11 | 31 | 42
  Asian | 3 | 1 | 4
  American Indian or Alaska Native | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Unknown | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 109 | 124 | 233

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Calcineurin Inhibitor-related Symptoms Severity Score
Description: The CIRS is a questionnaire that assesses five symptoms (from the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events [PRO-CTCAE]) that have been shown to be associated with calcineurin inhibitors. These symptoms include trembling hands, muscle cramps, muscle weakness, swollen gums, and increased hair growth. Each symptom is based on symptom severity in the last 7 days scaled from 0 (none) - 4 (very severe). The cumulative score ranges from 0-20, with higher scores indicating a worse outcome.
Time Frame: Baseline; 12 months
Population: 20 subjects in the Tacrolimus arm and 45 subjects in the Envarsus arm did not complete the CIRS questionnaire at the 12-month mark, therefore no data exists for those 65 subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tacrolimus Twice-daily | Envarsus XR
Number analyzed (Participants) | 88 | 72
score on a scale | -2.977 (14.053) | -3.139 (14.846)
Statistical Analysis 1: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Test type: Superiority; p = 0.944, t-test, 2 sided

2. Secondary Outcome: Change in the Severity Score in Each of the Five Individual CIRS Items
Description: The change in the severity score in each of the five individual CIRS items: trembling hands, muscle cramps, muscle weakness, swollen gums, and increased hair growth. The CIRS is a questionnaire that assesses five symptoms (from the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events [PRO-CTCAE]) that have been shown to be associated with calcineurin inhibitors. These symptoms include trembling hands, muscle cramps, muscle weakness, swollen gums, and increased hair growth. Each symptom is based on symptom severity in the last 7 days scaled from 0 (none) - 4 (very severe), with higher scores indicating a worse outcome.
Time Frame: Baseline; 12 months
Population: 20 subjects in the Tac arm and 45 subjects in the Envarsus arm didn't complete the CIRS questionnaire at the 12-month mark, therefore no data exists for those 65 subjects. 1 subject in the Tac arm and 1 in the Envarsus arm didn't complete the muscle weakness section of the questionnaire. 1 subject in the Tac arm didn't complete the swollen gums section of the questionnaire. 2 subjects in the Tac arm and 1 in the Envarsus arm didn't complete the hair growth section of the questionnaire.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Tacrolimus Twice-daily | Envarsus XR
Number analyzed (Participants) | 88 | 72
score on a scale
  Trembling Hands | 0 [-1 to 1] | 0 [-1 to 1]
  Muscle Cramps | 0 [0 to 0] | 0 [0 to 0]
  Muscle Weakness: number analyzed (Participants) | 87 | 71
  Muscle Weakness | 0 [-1 to 0] | 0 [-1 to 1]
  Swollen Gums: number analyzed (Participants) | 87 | 72
  Swollen Gums | 0 [0 to 0] | 0 [0 to 0]
  Increased Hair Growth: number analyzed (Participants) | 86 | 71
  Increased Hair Growth | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Trembling Hands; Test type: Superiority; p = 0.345, Kruskal-Wallis
Statistical Analysis 2: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Muscle Cramps; Test type: Superiority; p = 0.451, Kruskal-Wallis
Statistical Analysis 3: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Muscle Weakness; Test type: Superiority; p = 0.953, Kruskal-Wallis
Statistical Analysis 4: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Swollen Gums; Test type: Superiority; p = 0.579, Kruskal-Wallis
Statistical Analysis 5: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Increased Hair Growth; Test type: Superiority; p = 0.513, Kruskal-Wallis

3. Secondary Outcome: Number of Subjects With a Moderately Severe, Severe or Very Severe Score on Any CIRS Item
Description: Number of subjects in each treatment group with a moderately severe, severe or very severe score (2, 3 or 4) on any CIRS item. The CIRS is a questionnaire that assesses five symptoms (from the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events [PRO-CTCAE]) that have been shown to be associated with calcineurin inhibitors. These symptoms include trembling hands, muscle cramps, muscle weakness, swollen gums, and increased hair growth. Each symptom is based on symptom severity in the last 7 days scaled from 0 (none) - 4 (very severe). The cumulative score ranges from 0-20, with higher scores indicating a worse outcome.
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tacrolimus Twice-daily | Envarsus XR
Number analyzed (Participants) | 88 | 72
Participants | 18 | 28
Statistical Analysis 1: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Test type: Superiority; p = 0.010, Chi-squared

4. Secondary Outcome: Change in the Number of Subjects Who Had a Reduction in Severity of Calcineurin Inhibitor-related Symptoms
Description: The change in the number of subjects with a reduction in a CIRS item score from a severe or very severe score (3 to 4) to a mild to moderate (1 or 2) score from 4 months to 12 months.
Time Frame: 4 months; 12 months
Population: 29 subjects in the Tacrolimus arm and 54 subjects in the Envarsus arm did not complete the CIRS questionnaire at the 4-month mark, therefore no data exists for those 83 subjects. 2 subjects in the Tacrolimus arm only filled out a portion of the survey at the 4-month mark, due to this those two subjects were not included in the analysis for this outcome as a change in reduction of symptoms from very severe/severe to mild/moderate could not be calculated.
Measure: Count of Participants; unit: Participants
Arm/Group | Tacrolimus Twice-daily | Envarsus XR
Number analyzed (Participants) | 77 | 63
Participants | 8 | 8

5. Secondary Outcome: Change in the Number of Subjects Who Had at Least One Calcineurin Inhibitor-related Symptom Reduced by 1 Point or Greater
Description: The change in the number of subjects with a reduction in any single CIRS item by 1 point or greater from 4 months to 12 months.
Time Frame: 4 months; 12 months.
Population: 29 subjects in the Tacrolimus arm and 54 subjects in the Envarsus arm did not complete the CIRS questionnaire at the 4-month mark, therefore no data exists for those 83 subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Tacrolimus Twice-daily | Envarsus XR
Number analyzed (Participants) | 79 | 63
Participants | 43 | 30

6. Secondary Outcome: Transplant-related Symptoms as Measured by the Difference in Mean Transplant-related Symptoms (TRS) Score.
Description: The TRS is a 30-item questionnaire capturing 15 symptoms (from PRO-CTCAE) that have been shown to be associated with transplant and general health-related quality of life improvement. These symptoms include change in taste, constipation, diarrhea, swelling in arms or legs, palpitations, dry skin, darkening of skin, blurry vision, headache, insomnia, anxiety, sadness, discouraged, increase in appetite, and fatigue. Each symptom is based on symptom severity in the last 7 days and scaled from 0 (none) - 4 (very severe). Total scores range from 0 to 120, with higher scores indicating a worse outcome.
Time Frame: Baseline; 12 months
Population: 20 subjects in the Tacrolimus arm and 45 subjects in the Envarsus arm did not complete the TRS questionnaire at the 12-month mark, therefore no data exists for those 65 subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tacrolimus Twice-daily | Envarsus XR
Number analyzed (Participants) | 88 | 72
score on a scale | -1.375 (9.882) | -1.069 (8.421)
Statistical Analysis 1: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Test type: Superiority; p = 0.836, t-test, 2 sided

7. Secondary Outcome: Change in Health-related Quality of Life (HRQoL), as Measured by the Patient-Reported Outcomes Measurement Information System 29 (PROMIS-29) Health Profile.
Description: The PROMIS-29 questionnaire measures physical and mental health outcomes for patients. Patients responded to 29 questions in seven categories: physical function, pain interference, depressive symptoms, anxiety, ability to participate in social activities, and sleep disturbance. Scores were scaled so that an average healthy person would score 50 points. A higher score represents a worse outcome. Patient questionnaire responses are scored using the PROMIS-29 scoring algorithm. Scores were scaled to a mean of 50 for a healthy reference population with a standard deviation of 10.
Time Frame: Baseline; 12 months
Population: 36 subjects in the Tacrolimus arm and 56 subjects in the Envarsus arm did not complete the PROMIS-29 questionnaire at the 12-month mark, therefore no data exists for those 92 subjects.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Tacrolimus Twice-daily | Envarsus XR
Number analyzed (Participants) | 72 | 61
score on a scale | -10 [-22 to 1] | -20 [-32 to -5]
Statistical Analysis 1: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Test type: Superiority; p = 0.008, Kruskal-Wallis

8. Secondary Outcome: Change in Transplant-related Symptoms as Measured by the Difference in Transplant-related Symptoms (TRS) Score in for Each Individual Symptom
Description: The change in the transplant related symptoms score in each of the fifteen individual TRS items: change in taste, constipation, diarrhea, swelling in arms or legs, palpitations, dry skin, darkening of skin, blurry vision, headache, insomnia, anxiety, sadness, depression, increase in appetite, and fatigue. The TRS is a multi-item questionnaire capturing 15 symptoms (from PRO-CTCAE) that have been shown to be associated with transplant and general health-related quality of life improvement. These symptoms include change in taste, constipation, diarrhea, swelling in arms or legs, palpitations, dry skin, darkening of skin, blurry vision, headache, insomnia, anxiety, sadness, depression, increase in appetite, and fatigue. Each symptom is based on symptom severity in the last 7 days and scaled from 0 (none) - 4 (very severe), with higher scores indicating a worse outcome.
Time Frame: Baseline; 12 months
Population: 20 in Tac arm,45 in XR arm didn't complete TRS at 12months,therefore no data exists for the 65 subjects.1 in XR arm didn't complete taste/palpitation/headache/insomnia/fatigue sections.1 in Tac arm didn't complete appetite/swelling/palpitation/fatigue/anxiety/depression section.3 in XR arm didn't complete diarrhea/depression/sadness sections.2 in Tac arm didn't complete vision/sadness sections.3 in Tac arm didn't complete headache section.8 in Tac arm,7 in XR arm didn't complete darkskin section
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Tacrolimus Twice-daily | Envarsus XR
Number analyzed (Participants) | 88 | 72
score on a scale
  Taste Change: number analyzed (Participants) | 88 | 71
  Taste Change | 0 [0 to 0] | 0 [-1 to 0]
  Appetite: number analyzed (Participants) | 87 | 72
  Appetite | 0 [0 to 0] | 0 [-1 to 1]
  Constipation | 0 [-1 to 0] | 0 [-1 to 0]
  Diarrhea: number analyzed (Participants) | 88 | 69
  Diarrhea | 0 [-1 to 0] | 0 [-1 to 0]
  Swelling: number analyzed (Participants) | 87 | 72
  Swelling | 0 [0 to 0] | 0 [-2 to 1]
  Palpitations: number analyzed (Participants) | 87 | 71
  Palpitations | 0 [0 to 0] | 0 [-2 to 0]
  Dry Skin | 0 [-1 to 0] | 0 [-1 to 0]
  Darker Skin: number analyzed (Participants) | 80 | 65
  Darker Skin | 0 [0 to 0] | 0 [0 to 0]
  Blurry Vision: number analyzed (Participants) | 86 | 72
  Blurry Vision | 0 [0 to 0] | 0 [0 to 0]
  Headache: number analyzed (Participants) | 85 | 71
  Headache | 0 [-1 to 1] | 0 [-1 to 2]
  Insomnia: number analyzed (Participants) | 88 | 71
  Insomnia | -1 [-2 to 0] | 0 [-2 to 1]
  Fatigue: number analyzed (Participants) | 87 | 71
  Fatigue | -1 [-2 to 0] | -1 [-2 to 0]
  Anxiety: number analyzed (Participants) | 87 | 72
  Anxiety | 0 [0 to 0] | 0 [-2 to 0]
  Depression: number analyzed (Participants) | 87 | 69
  Depression | 0 [0 to 0] | 0 [0 to 0]
  Sadness: number analyzed (Participants) | 86 | 69
  Sadness | 0 [0 to 0] | 0 [0 to 1]
Statistical Analysis 1: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Taste Change; Test type: Superiority; p = 0.314, Kruskal-Wallis
Statistical Analysis 2: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Appetite; Test type: Superiority; p = 0.486, Kruskal-Wallis
Statistical Analysis 3: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Constipation; Test type: Superiority; p = 0.452, Kruskal-Wallis
Statistical Analysis 4: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Diarrhea; Test type: Superiority; p = 0.750, Kruskal-Wallis
Statistical Analysis 5: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Swelling; Test type: Superiority; p = 0.764, Kruskal-Wallis
Statistical Analysis 6: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Palpitations; Test type: Superiority; p = 0.726, Kruskal-Wallis
Statistical Analysis 7: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Dry Skin; Test type: Superiority; p = 0.421, Kruskal-Wallis
Statistical Analysis 8: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Darker Skin; Test type: Superiority; p = 0.679, Kruskal-Wallis
Statistical Analysis 9: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Blurry Vision; Test type: Superiority; p = 0.779, Kruskal-Wallis
Statistical Analysis 10: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Headache; Test type: Superiority; p = 0.533, Kruskal-Wallis
Statistical Analysis 11: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Insomnia; Test type: Superiority; p = 0.668, Kruskal-Wallis
Statistical Analysis 12: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Fatigue; Test type: Superiority; p = 1.00, Kruskal-Wallis
Statistical Analysis 13: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Anxiety; Test type: Superiority; p = 0.232, Kruskal-Wallis
Statistical Analysis 14: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Depression; Test type: Superiority; p = 0.566, Kruskal-Wallis
Statistical Analysis 15: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Sadness; Test type: Superiority; p = 0.038, Kruskal-Wallis

9. Secondary Outcome: Change in Overall Tolerability or Patient Bother Due to Side Effects
Description: Measured by item GP5 ("I am bothered by side effects of treatment") from the FACT-G Questionnaire. FACT-G GP5 is a single-item measure from the Functional Assessment of Cancer Therapy (FACT) scale, specifically designed to assess patient-reported tolerability to cancer treatments. Subjects are asked to rate their level of tolerability on a scale of 0 (not at all bothered) to 4 (very much bothered), with a higher score indicating a worse outcome.
Time Frame: Baseline; 12 months
Population: 21 subjects in the Tacrolimus arm and 45 subjects in the Envarsus arm did not complete the FACT-G questionnaire at the 12-month mark, therefore no data exists for those 66 subjects.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Tacrolimus Twice-daily | Envarsus XR
Number analyzed (Participants) | 87 | 72
score on a scale | 0 [-1 to 0] | 0 [-1 to 0]
Statistical Analysis 1: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Test type: Superiority; p = 0.754, Kruskal-Wallis

10. Secondary Outcome: Change in Medication Adherence
Description: Defined as the percentage of prescribed doses taken each day
Time Frame: 12 months
Population: Data for this outcome measure were not collected in either treatment arm. The electronic data capture system was configured incorrectly and did not include the fields required to record medication adherence. As a result, the study team was unable to collect adherence data for any participants.
Arm/Group | Tacrolimus Twice-daily | Envarsus XR
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in Patient Medication Satisfaction as Assessed by Question 14 of the Treatment Satisfaction Questionnaire for Medication.
Description: Question 14 of the Treatment Satisfaction Questionnaire for Medication measures medication satisfaction on a 7-item scale ranging from 0 (Extremely Dissatisfied) to 7 (Extremely Satisfied), with higher scores indicating better satisfaction.
Time Frame: Baseline; 12 months
Population: 99 subjects in the Tacrolimus arm and 116 subjects in the Envarsus arm did not complete the Treatment Satisfaction questionnaire at the 12-month mark, therefore no data exists for those 215 subjects.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Tacrolimus Twice-daily | Envarsus XR
Number analyzed (Participants) | 9 | 1
score on a scale | 0 [-1 to 1] | 1 [1 to 1]
Statistical Analysis 1: Comparison: Tacrolimus Twice-daily vs Envarsus XR; Test type: Superiority; p = 0.371, Kruskal-Wallis

12. Secondary Outcome: Correlation Between de Novo DSA and Degree of Taking and Timing Adherence
Description: Proportion of patients at different adherence thresholds of taking and timing adherences between 4 months and 12 months post transplant will be correlated with the presence or absence of dnDSA by 12 months post-transplant
Time Frame: 4 months; 12 months
Population: Data for this outcome measure were not collected in either treatment arm. The electronic data capture system was configured incorrectly and did not include the fields required to record correlation between de novo DSA and degree of taking and timing adherence. As a result, the study team was unable to collect correlation between de novo DSA and degree of taking and timing adherence data on any participant.
Arm/Group | Tacrolimus Twice-daily | Envarsus XR
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Adverse Events
Description: Number of adverse events reported
Time Frame: 12 months
Measure: Number; unit: events
Arm/Group | Tacrolimus Twice-daily | Envarsus XR
Number analyzed (Participants) | 109 | 124
events | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through study completion, approximately 12 months.
Description: Adverse events were collected through monthly blood labs and safety assessments.
Arm/Group | Tacrolimus Twice-daily | Envarsus XR
All-Cause Mortality (participants affected / at risk) | 1/109 | 3/124
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/124
Other Adverse Events (participants affected / at risk) | 0/109 | 0/124

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT03979365/Prot_SAP_000.pdf